CLINICAL TRIAL: NCT05766644
Title: Open-label, Randomized Comparative Clinical Trial on the Clinical Effect of App-based Education Program in Patients With Chronic Kidney Disease
Brief Title: App-based Education Program for CKD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Inje University (Other)
Collaborators: Hallym University Kangnam Sacred Heart Hospital (Other); KangWon National University Hospital (Other); Korea University Guro Hospital (Other); Korea University Ansan Hospital (Other); Seoul National University (Other); Ministry of Health & Welfare, Korea (Other Government)
Responsible Party: Principal Investigator, Hoseok Koo, Director, Inje University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Beans_CKD Education 1.0
Record Dates: First submitted 2023-02-27; First posted 2023-03-13 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Renal Insufficiency, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Educational Status

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Usual care, with no guide on app use. Surveys are administered via Short Message Services links.
- Education (Experimental): Enrolled in a mobile app-based education program, with guidance from a healthcare professional. All educational materials and surveys are provided via the app.
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — An 8-week program providing educational materials via a mobile app for chronic kidney disease management. Materials consist of videos, card news, and live online seminars with a Q&A session. Topics are on general disease information, nutrition, and exercise.
  Arms: Education

SUMMARY:
A randomized control trial to test the effect of a mobile app-based educational program for Chronic Kidney Disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with CKD Stage 1~5
* Have been receiving CKD treatment for more than 6 months
* Owns an android mobile phone

Exclusion Criteria:

* Diagnosed with cancer within 5 years of recruitment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-10-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (SF-36v2) | 48 days
  36-Item Short Form Health Survey, version 2. Scores range from 0 to 100, higher value corresponding to better outcome (better quality of life)
MIS | 55 days
  10-item nutritional status measured with Malnutrition Inflammation Score. Scores range from 0 to 30, higher value corresponding to worse outcome (higher risk of malnutrition)
Potassium | 56 days
  Serum potassium levels obtained from routine blood test.
Phosphate | 56 days
  Serum phosphate levels obtained from routine blood test.
Albumin | 56 days
  Serum albumin levels obtained from routine blood test.

SECONDARY OUTCOMES:
Depression | 55 days
  21-item depression score measured with Korean-Beck Depression Inventory. Scores range from 0 to 63, higher value corresponding to worse outcome (severe depression).
Insomnia | 48 days
  7-item insomnia score measured with Insomnia Severity Index in Korean. Scores range from 0 to 28, higher value corresponding to worse outcome (severe insomnia)
Sodium intake behavior | 0 days
  15-item sodium intake behavior score. Scores range from 0 to 15, higher values corresponding to worse outcome (higher tendency to prefer salty food).
Sodium intake attitude | 0 days
  17-item sodium intake attitude score. Scores range from 0 to 17, higher values correspond ing to better outcome (more willing to reduce sodium intake).
Creatinine | 56 days
  Creatinine levels obtained from routine blood test.

CONTACTS AND LOCATIONS:
Overall Officials: Hoseok Koo, Principal Investigator — Inje University
Locations (1):
- Inje University Seoul Paik Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No